CLINICAL TRIAL: NCT04066751
Title: A Multicenter Randomized, Double-blind, Phase 2, Placebo Controlled Study to Determine the Safety and Efficacy of Ivacaftor (VX-770) for the Treatment of Chronic Obstructive Pulmonary Disease (The Multicenter Topic Trial)
Brief Title: The Multicenter Topic Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started due to change in availability of study drug
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Mark Dransfield, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300003967; P30DK072482 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivacaftor (Active Comparator): Ivacaftor, 150 mg PO every 12 hrs for 84 days
  Interventions: Drug: Ivacaftor
- Placebo (Placebo Comparator): Placebo, 150 mg PO every 12 hrs for 84 days
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — Ivacaftor will be supplied as a tablet for oral administration, film-coated, 150 mg
  Other Names: Kalydeco

SUMMARY:
The purpose of this protocol is to test the safety, pharmacokinetics, and pharmacodynamics of the Cystic fibrosis transmembrane conductance regulator (CFTR) potentiator, ivacaftor in patients with chronic obstructive pulmonary disease (COPD) and chronic bronchitis. This project will investigate the hypothesis that ivacaftor can augment CFTR activity in individuals with COPD who exhibit chronic bronchitis, resulting in meaningful improvements in epithelial function and respiratory health. The study is a multicenter, randomized, double-blind, placebo-controlled, stratified study of orally-administered ivacaftor.

DETAILED DESCRIPTION:
Like CF, COPD is characterized by small airway mucus obstruction that is associated with accelerated loss of lung function and mortality. Our preliminary data indicate that cigarette smoke exerts deleterious effects on airway epithelial function including the reduction of CFTR activity, enhanced mucus expression, and a pronounced reduction in mucociliary transport (MCT). Preliminary data also indicate that approximately 50% of patients with COPD have reduced CFTR activity, as detected in the upper airways, lower airways, and sweat glands. Furthermore, CFTR dysfunction is independently associated with chronic bronchitis, can persist despite smoking cessation, and can be reversed by the CFTR potentiator ivacaftor (VX-770) in vitro by activating wild-type CFTR, resulting in a robust increase in MCT. Combined with unprecedented clinical improvement via augmented mucociliary clearance in CF patients with a responsive CFTR mutation treated with ivacaftor, these data indicate that CFTR represents a viable therapeutic target to address mucus stasis in a large subset of COPD patients (potentially representing over 4 million patients in the U.S. alone). This project will investigate the hypothesis that ivacaftor can augment CFTR activity in individuals with COPD who exhibit chronic bronchitis, resulting in meaningful improvements in epithelial function and respiratory health. Our initial pilot study in patients with COPD and chronic bronchitis demonstrated that ivacaftor was safe, demonstrated stable pharmacokinetics, and exhibited a trend towards efficacy in patient-reported outcomes (PROs) and sweat chloride. The current trial will test the safety, pharmacokinetics, and pharmacodynamics of ivacaftor in a larger number of COPD patients with chronic bronchitis and for a longer treatment period, evaluating the potential of CFTR potentiator therapy to address acquired CFTR dysfunction in this population and set the stage for larger and longer-term trials in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 40-80
* A Clinical diagnosis of COPD as defined by GOLD
* At Least a 10 pack year smoking history
* Exhibit symptoms of chronic bronchitis as defined by the Medical Research Council
* FEV1% predicted ≥ 35% and ≤80% Post Bronchodilator
* Clinically stable in the last 4 weeks with no evidence of COPD exacerbation
* Weight of 40 kg-120 kg
* Willingness to use at least one form of acceptable birth control including abstinence, condom with spermicide, or hormonal contraceptives from time of signing ICF through study follow up visit
* Willing to monitor blood glucose if known history of insulin dependent diabetes mellitus
* Capable of giving signed informed consent

Exclusion Criteria:

* Current Diagnosis of Asthma
* Known Diagnosis of Cystic Fibrosis
* Use of Continuous Oxygen Therapy of greater than 2 liters per minute - patients on 2 liters of Oxygen or less will be excluded if they have been hospitalized for COPD in the prior year or had more than 2 exacerbations requiring steroids and/or antibiotics in the prior year.
* Documented history of drug abuse within the last year
* Subjects should not have a pulmonary exacerbation or changes in therapy for pulmonary disease within 28 days before receiving the first dose of study drug.
* Cirrhosis or elevated liver transaminases > 3X ULN
* GFR < 50 estimated by Cockroft-Gault
* Any illness or abnormal lab finding that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Pregnant or Breastfeeding
* Subjects taking moderate or strong inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit juice. (Excluded medications and foods including the drugs and foods listed in the IRB HSP application.)
* Uncontrolled Diabetes
* Recent (e.g 1year) arterial thrombotic events (peripheral arterial disease, thrombotic stroke)
* Clinically significant arrhythmias requiring anti-arrhythmic agent(s) or conduction abnormalities that in the opinion of the investigator affect patient safety
* A standard digital ECG demonstrating QTc >450 msec for men and > QTc 470 msec for women at screening. If QTc exceeds 450 msec for men and > QTc 470 msec for women at the screening ECG, the ECG should be repeated 2 more times during the screening period, and the subject will be excluded if the average of the 3 QTc values is >450 msec for men and > QTc 470 msec for women.
* Angina symptoms
* History of MI or revascularization procedure within the last three years prior to screening
* Clinically significant congestive heart failure (known LVEF <= 45%, cor pulmonale, diastolic heart failure, etc)
* Patients with stable coronary artery disease are eligible
* History of stroke/CVA or non-skin cancer <5 years prior

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
CFTR activity | assessed at day1, day 28, day 56, and day 84
  Change in peripheral CFTR activity as detected by sweat chloride testing
FEV1 | assesed at day 1, day 28, day 56, and day 84
  Change in lung function as measured by FEV1 (Pulmonary Function testing.)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dransfield, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No